CLINICAL TRIAL: NCT05194774
Title: Outcomes of The Greater Trochanter Epiphysiodesis In Treatment Of Children With Hip Pathology
Brief Title: Greater Trochanter Epiphysiodesis In Hip Pathology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Muhammed Yasser, principal investigator, Al-Azhar University
Other Study IDs: GTE
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GT overgrowth group: pediatric patients with greater trochanter overgrowth
  Interventions: Procedure: Greater Trochanter epiphysiodesis

INTERVENTIONS:
Procedure: Greater Trochanter epiphysiodesis — epiphysiodesis by cortical screw and washer

SUMMARY:
One of the most common problems in the treatment of pediatric patients with various disorders of the hip joint is the formation of deformity of the proximal femur, such as abnormal growth of the greater trochanter, which causes it to be positioned high in relation to the femoral head. This condition is called "relative overgrowth of the greater trochanter" (ROGT).

ELIGIBILITY:
Inclusion Criteria:

* emerging deformities of the proximal femur with a high position of the greater trochanter, in which its apex was located above the center of the femoral head but below its superior pole; changes in the structure of the femoral neck, accompanied by its shortening; functioning growth zone of the greater trochanter at the time of intervention; and patients without surgical treatment history

Exclusion Criteria:

* hip dislocation upon examination; patients with varus deformity of the femoral neck (neck-shaft angle <120°), patients with complications of surgical interventions, trauma, rickets, and rheumatoid arthritis; and patients with neurological disorders and Refusal to participate in this study

Ages: 5 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: The patients come to the outpatient clinic and underwent clinical and radiological examination will be done , then preparation to surgery by screw
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Radiological measurments | 12 month
  articulo-trochanteric distance

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCarthy JJ, Weiner DS. Greater trochanteric epiphysiodesis. Int Orthop. 2008 Aug;32(4):531-4. doi: 10.1007/s00264-007-0346-5. Epub 2007 Mar 10. PMID 17351775